CLINICAL TRIAL: NCT04935489
Title: Accelerated Intermittent Theta Burst Stimulation for Depressed Patients During the Covid-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Shores Centre for Mental Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Robyn Waxman, Head of Brain Stimulation Clinic, Ontario Shores Centre for Mental Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-008-B
Record Dates: First submitted 2021-06-11; First posted 2021-06-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients receiving accelerated rTMS (Experimental)
  Interventions: Device: Intermittent Theta Burst Stimulation (form of repetitive transcranial magnetic stimulation) given in an accelerated form

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation (form of repetitive transcranial magnetic stimulation) given in an accelerated form — The intervention is used regularly for patients with treatment resistant depression, however, in this trial it will be given multiple times per day and over less days than the usual protocol

SUMMARY:
Repetitive Transcranial Magnetic Stimulation (rTMS) using intermittent theta burst stimulation (iTBS) has been found to be a non inferior protocol to standard rTMS for the treatment of major depressive disorder. An accelerated course is of particular interest given the safety profile of the procedure and the potential to treat people more quickly making the treatment more accessible. This study aims to assess the feasibility and clinical outcomes of a high dose iTBS protocol in patients with depression in the context of unipolar or bipolar II disorder who are waiting for Electroconvulsive therapy (ECT) or rTMS due to degree of treatment resistance or severity of symptoms. This is a prospective, open-label, interventional pilot study wherein patients who have been diagnosed with major depressive disorder and referred to brain stimulation clinic, will be recruited for the treatment. Patients will be administered eight questionnaires before and after the treatment to assess the change in clinical outcomes.

DETAILED DESCRIPTION:
Participants will receive same stimulation protocol, however they will be given 6 times per day instead of once per day. Each Treatment will consist of a single iTBS treatment delivering 600 puses of iTBS (bursts of 3 pulses at 50 Hz, bursts repeated at 5 Hz, with a duy cycle of 2 seconds on, 8 seconds off, over 60 cycles and it takes about 3 minutes at a target of 90 to 120% of the subject's resting motor threshold. Treatment will be given through the device that is usually used, which is Magpro by Magventure, B70 Fluid-Cooled Coil .

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Unipolar Depression or Bipolar II depression based on the MINI - no psychotic features
* Pass the TMS safety screen on the brain stimulation consultation template Voluntary and Competent to consent to treatment

Exclusion Criteria:

* Have a MINI confirmed diagnosis of a substance use disorder within the last month
* Have a concomitant major unstable medical illness, cardiac pacemaker or implanted mediation pump
* Have a lifetime MINI diagnosis of bipolar I, or schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder.
* Have any significant neurological disorder or insult including but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT, or a febrile seizure of infancy or single seizure related to a known drug related event, cerebral aneurysm, or significant head trauma with loss of consciousness for greater than 5 minutes
* Have an intracranial implant (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head (excluding the mouth) that cannot be safely removed.
* Currently taking more than lorazepam 2mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit rTMS efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Remission of depressive symptoms using the Hamilton Depression Rating Scale (HAM - D or HDRS) - 17 version | at screening (within a week of starting treatment) to a week post treatment
  Severity of depressive symptoms being measured pre and post treatment - remission is less than 8 (low score is less depression, higher score - more depressive symptoms, range is 0 to 53)

SECONDARY OUTCOMES:
Response to treatment with reduction of 50% in depressive symptoms on HAM-D - 17 and PHQ - 9 (patient health questionnaire) | at screening (within a week of starting treatment) to a week post treatment
  Change in severity of depressive symptoms (same as primary outcome description)
Response of anxiety symptoms - reduction by 50% - Generalized Anxiety disorder scale (GAD-&) | at screening (within a week of starting treatment) to a week post treatment
  Change in severity of anxiety symptoms - higher the score, more anxiety symptoms, range 0 to 21
Change in World Health Organization Disability assessment scale (WHODAS) | at screening (within a week of starting treatment) to a week post treatment
  severity of disability ( 40 to 180 - higher score = more disabled)
Change in the Quality of Life, Enjoyment, and Satisfaction Questionnaire (QUAL-ES-Q) | at screening (within a week of starting treatment) to a week post treatment
  Change in rated quality of life, score range from 14 to 70 ( higher score = better quality of life)
Improvement overall using the Clinical Global Severity/Impression Scale (CGI-I) | at screening (within a week of starting treatment) to a week post treatment
  Change in severity of illness (1 - much worse, 7 - most improved)
Patient Health Questionnaire (PHQ-9) - Response to symptoms | at screening (within a week of starting treatment ) to a week post treatment
  reduction in depression score by 50% - higher the score - more depressive symptoms, scored from 0 to 27

OTHER OUTCOMES:
Adverse effects of the treatment | during and after each rTMS treatment during acute treatment and up to a week after treatment
  Looking at occurrence of adverse effects - screened during/after each treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Waxman, Principal Investigator — Ontario Shores
Locations (1):
- Robyn, Whitby, Ontario, Canada